CLINICAL TRIAL: NCT01826383
Title: Improving Parental Soothing by Video: A Randomized Controlled Trial
Brief Title: Improving Parental Soothing by Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, RRiddell, Associate Professor, York University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: York HPRC 2013-004
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Acute Pain
Keywords: Infant; Immunization
MeSH Terms: conditions — Acute Pain | interventions — Exergaming

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Video (Experimental): This is a five-minute video that coaches parents about how to soothe their infant post-immunization.
  Interventions: Behavioral: Active-Video
- Placebo Video (Placebo Comparator): This is a video identical to that of the active video, except no specific instructions regarding how to soothe an infant post-immunization are given.
  Interventions: Behavioral: Placebo Video

INTERVENTIONS:
Behavioral: Active-Video — This group will watch an active-video with pain management strategies for parents
  Arms: Active Video
Behavioral: Placebo Video — This group will watch a placebo-video describing immunization generally.
  Arms: Placebo Video

SUMMARY:
This study sets out to compare the effectiveness of a parent pain management coaching video that is 5-minutes in length. The investigators will be comparing an active-video to a placebo-video of equal length (and identical formatting). Participants will be 6 or 18 month infants undergoing routine immunization. The investigators hypothesize the active video will result in a lowering of infant pain expressed post-immunization (3 minutes) and the increase in the parental use of distraction, physical comfort, and rocking.

DETAILED DESCRIPTION:
Our goal is to determine if a video instructing parents on the principles of soothing their infant following immunization will influence soothing behaviours exhibited by parents, and pain reactivity and regulation in infants. We plan to present parents of young infants (6 months) and older infants (18 months) with either a Treatment Video instructing them on the ABCD's (Assess Anxiety, Belly Breathe, Calm Close Cuddle, Distraction; Copyright R. Pillai Riddell) of pain management or a Placebo Video with neutral information. There is very minimal risk because our suggestions are based on what parents deemed 'sensitive' (in our ongoing longitudinal study) were doing naturally i.e., without any intervention in their day-to-day lives. Additionally, in a separate study, that already received ethics approval, parents viewed these videos without any negative side effects.

Participants will be adult parents from one of two clinics in the Greater Toronto Area who bring their infant in for a routine immunization (12 or 18 months). In our cohort study (where we simply videotape dyads in the clinic).

Parents will be asked to complete a brief questionnaire (Parent Information Sheet) entailing basic demographic information and preimmunization ratings of their worry about their infant's pain from the immunization. The parents will also be asked to complete the 18-item Brief Symptom Inventory (BSI-18) and the Negative Affect subscale (IBQ-R Very short form), in addition to demographic information. The parents will subsquently be asked to view a brief video (Treatment or Placebo Video) discussing the ABCD's of pain management described above. During the infant's routine immunization procedure the parents and infant will be videotaped for approximately 10 minutes, and the parent will be asked a few brief questions post immunization including ratings of their infant's pain from the immunization procedure and the helpfulness of the video.

ELIGIBILITY:
Inclusion Criteria:

* Infants must be 6 or 18 months old receiving a routine immunization injection.
* Parents must be fluent in English.
* Only one child per family can be enrolled.

Exclusion Criteria:

* No suspected developmental delays or chronic illnesses.
* Time spent in a Neonatal Intensive Care Unit.
* Born more than 3 weeks premature.

Ages: 5 Months to 20 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Modified Behaviour Pain Scale | 3 minutes post-last needle
  Infant pain regulation was operationalized using The Modified Behaviour Pain Scale (MBPS), modified by Taddio et al. (1995) for use with infants during office procedures. The measure rates the severity of distress reflected in three types of infant pain behaviours: (1) facial expressions; (2) cry; and (3) body movements during 15-second epochs post-immunization (for 3 minutes). Infants are assigned a score from 0 to 3 (or 0 to 4 on the cry scale), with larger values indicating a more intense behavioural response (Total Range 0-10)

SECONDARY OUTCOMES:
Measure of Adult and Infant Soothing and Distress | 3 minutes post-last needle
  The MAISD (Measure of Adult and Infant Soothing and Distress; Cohen et al., 2005) is a behavior observation scale that was developed to examine the discrete behaviors exhibited by parents during children's invasive medical procedures. Rather than attempting to examine all behaviors, only those that were viewed as being potentially impacted by the treatment video will be included. Thus, distraction, rocking, physical comfort were selected. Each behaviour is coded every 5 seconds for either presence or absence (0 or 1). Three separate scores will be derived for each behaviour (distraction, rocking, physical comfort).

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca R Pillai Riddell, PhD, Principal Investigator — York University
Locations (2):
- Canada (2):
  - Dr. Saul Greenberg's Pediatric Clinic, Toronto, Ontario
  - Dr. Hartley Garfield's Pediatric Clinic, Toronto, Ontario

REFERENCES:
- [Background] Taddio A, Nulman I, Koren BS, Stevens B, Koren G. A revised measure of acute pain in infants. J Pain Symptom Manage. 1995 Aug;10(6):456-63. doi: 10.1016/0885-3924(95)00058-7. PMID 7561228
- [Background] Cohen, L.L., Bernard, R., McClellan, C., MacLaren, J. (2005). Assessing Medical Room Behaviour During Infants' Painful Procedures: The Measure of Adult and Infant Soothing and Distress (MAISD). Children's Health Care., 34, p. 81-94.